CLINICAL TRIAL: NCT05558358
Title: Deep Brain Stimulation (DBS) for Methamphetamine Use Disorder
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 18-0254; UG3DA054746 (NIH)
Record Dates: First submitted 2022-09-19; First posted 2022-09-28 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Methamphetamine Use Disorder

STUDY DESIGN:
Intervention Model Description: All participants undergo surgery. Some receive 6 months of active DBS stimulation of the bilateral nucleus accumbens followed by 6 months of sham stimulation. While some receive the opposite order.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and all study personnel are blinded to subject assignment except the physician completing DBS programming.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 1 (Experimental): Randomized sham-controlled crossover design - participants have baseline assessments/evaluation, 1 week detoxification, surgery, 30 days residential care, then begin DBS stimulation, 12 weeks IOP/CM and are followed for 52 weeks.
  Interventions: Device: Experimental 1 - DBS of bilateral NAc - 6 months of active stimulation -- > 6 months of sham stimulation
- 2 (Experimental): Randomized sham-controlled crossover design - participants have baseline assessments/evaluation, 1 week detoxification, surgery, 30 days residential care, then begin DBS stimulation, 12 weeks IOP/CM and are followed for 52 weeks.
  Interventions: Device: Experimental 2 - DBS of bilateral NAc - 6 months of sham stimulation -- > 6 months of active stimulation

INTERVENTIONS:
Device: Experimental 1 - DBS of bilateral NAc - 6 months of active stimulation -- > 6 months of sham stimulation — 6 months of active stimulation -- > 6 months of sham stimulation
  Arms: 1
Device: Experimental 2 - DBS of bilateral NAc - 6 months of sham stimulation -- > 6 months of active stimulation — 6 months of sham stimulation -- > 6 months of active stimulation
  Arms: 2

SUMMARY:
We will evaluate the effects of deep brain stimulation (DBS) of bilateral nucleus accumbens (NAc) added to background treatment for treatment refractory Methamphetamine Use Disorder (MUD). This is a small randomized cross-over study to demonstrate feasibility and safety, test treatment outcomes (use, craving), and identify novel biological targets (NAc local field potentials (LFP) and functional MRI).

DETAILED DESCRIPTION:
In a randomized cross-over design of DBS of the nucleus accumbens (NAc) for treatment refractory methamphetamine use disorder (MUD, n=5), we will test safety, feasibility, effect on clinical outcomes (craving and use), and seek to identify biological targets (using cue craving during recording of local field potentials and MRI).

ELIGIBILITY:
Inclusion Criteria:

Adults (men and non-pregnant or nursing women) between 22-65 years of age will be eligible for enrollment, if meeting the following criteria:

1. Current diagnosis of DSM-5 MUD (with past year specifier of severe and at least a 5-year history);
2. Failed at least 2 prior treatment episodes (defined as outpatient or inpatient, utilizing a previously validated psychosocial treatment for addiction such as cognitive behavioral therapy, contingency management, motivational interviewing (Stuart et al., 2019) and not counting episodes with only detoxification) for MUD, with at least 1 episode having been residential;
3. Provides a urine drug screen positive for mAMP;
4. Endorses at least 10 days of mAMP use in the past month;
5. Able to complete 1 week of inpatient detoxification prior to surgery and 4 weeks of inpatient treatment following surgery;
6. No change in current psychiatric medication regimen, or medication free, for at least 4 weeks prior to entry;
7. Able to provide informed consent;
8. Able to comply with all testing and follow-up requirements as defined by study protocol (including providing a home address and two local collateral contacts);
9. Medically able to undergo DBS procedure as assessed by Study Neurosurgeon;
10. Has platelet count, PT and PTT within normal laboratory limits;
11. Adequate English proficiency for study consent, and completion of the study instruments;
12. Reside in the state of Colorado.

Exclusion Criteria:

1. Lifetime non-substance-induced psychotic disorders, schizophrenia, or schizoaffective disorder defined by DSM-5;
2. Current diagnosis of DSM-5 drug use disorder other than stimulant, alcohol, cannabis or nicotine use disorder;
3. Non-substance-induced manic episode within the past 3 years or major depressive episode in the past year;
4. Current clinically significant neurological disorder or medical illness;
5. Presence of a clinically significant abnormality on preoperative MRI;
6. Inability to have an MRI;
7. Inability to undergo general anesthesia required for tunneling of extension cable and placement of the batteries;
8. Pregnancy or lack of use of effective contraception in women of childbearing age, as assessed by urine pregnancy test and self-report (participants will consent to continue effective contraceptives during the study);
9. Coagulopathy, as determined by PT, PTT, platelet count, and medical history;
10. History of recurrent infections;
11. Inability to adhere to the requirements of the study;
12. Imminent risk of suicide as determined by Study Psychiatrist's assessment and investigators' clinical judgment or past-year suicide attempt, any positive response on baseline Columbia Suicide Severity Scale or history of parental completed suicide;
13. Active criminal justice involvement (i.e., any unresolved legal problems that could jeopardize continuation or completion of the study);
14. History of head injury with loss of consciousness for more than 15 minutes, neurological illness (including primary seizure disorder);
15. Diagnosis of dementia;
16. Conditions requiring diathermy.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of study-emergent adverse events | 56 weeks
  Participants will be closely monitored for adverse events throughout the study including regular meetings with study staff and administration of the COMBINE SAFTEE during each programming session.

SECONDARY OUTCOMES:
Methamphetamine use | Measured during weeks 26-30 and weeks 52-56 (last month on stimulation and sham)
  Operationalized as the highest number of consecutive days of no methamphetamine use in the final month of sham vs. final month of active stimulation.
Methamphetamine use | Measured during weeks 26-30 and weeks 52-56 (last month on stimulation and sham)
  Operationalized as the number of days methamphetamine is used in the final month of sham vs. final month of active stimulation.
Methamphetamine craving | Comparing weeks 26-30 and weeks 52-56
  Measured weekly using the Stimulant Craving Questionnaire-Brief where each item is scored 0-6 (from Strongly Disagree=0 to Strongly Agree=6) with items #4 and #7 reverse scored. We will average all 10 items as the total score, with higher scores indicating greater levels of craving in the final month of sham vs. final month of active stimulation.
Local Field Potential | baseline through week 56
  Electrophysiologic data - three types of LFP data that will be collected: (a.1) BrainSense™ Streaming assessed in the laboratory during the cue-craving task at baseline, 6, and 12 months; (a.2) BrainSense™ Events will be triggered by the participant using the patient programmer when he/she experiences craving; (a.3) BrainSense™Timeline records 10 minute averages of power spectral data within a 5 Hz window throughout the 12 month UG3 trial.
MRI | 56 weeks
  Cue craving MRI data will be collected at baseline, week 30 and week 56
MRI | 56 weeks
  Resting state MRI data will be collected at baseline, week 30 and week 56
Behavioral Inhibition System/Behavioral Approach System (BIS/BAS) | 56 weeks
  BIS/BAS will be collected at baseline, week 30 and week 56 Behavioral inhibition system score, assessing tendency to withdraw from aversive conditioned stimuli, and a behavioral activation score assessing tendency to approach appetitive stimuli.
  This is a 24-item scale with all items rated on a 4 point scale. With appropriate reverse scoring, this will be used to create BIS score (items 2, 8, 13, 16, 19, 22, 24), BAS Drive (items 3, 9, 12, 21), BAS Fun Seeking (5, 10, 15, 20) and BAS Reward Responsiveness (items 4, 7, 14, 18, 23) scores.
Impulsiveness | 56 weeks
  Barratt Impulsiveness Scale (BIS-11) will be collected at baseline, week 30 and week 56 This 30 item measure questionnaire (using a 1-4 scale for each item) generates a total score, along with Attentional, Motor and Nonplanning second order factors.
Sensation seeking | 56 weeks
  This 40-item questionnaire, measured at baseline, week 30 and week 56, provides, with appropriate reverse scoring, a total score (items 1-40), and 4 subscales: Disinhibition (1, 12, 13, 25, 29, 30, 32, 35, 36), Boredom Susceptibility (2, 5, 7, 8, 15, 24, 27, 31, 34, 39), Thrill and Adventure Seeking (3, 11, 16, 17, 20, 21, 23, 28, 38, 40) and Experience Seeking (4, 6, 9, 10, 14, 18, 19, 22, 26, 37).
Anhedonia | 56 weeks
  The Snaith-Hamilton Pleasure Scale, measured at baseline, week 30 and week 56, is a 14 item questionnaire (all rated on a 4 point Likert scale) and covers four domains of hedonic experience (interest/pastimes, social interaction, sensory experience and food/drink). With appropriate reverse scoring, we will use total score.
Delay Discounting | 56 weeks
  The MCQ, measured at baseline, week 30 and week 56, is a 27 item self administered questionnaire that examines delay discounting and can be hand scored using available tables. We will use the mean of the k at indifference between 2 questions that reflect a change between choosing a delayed vs. immediate reward.
Risk taking | 56 weeks
  Balloon Analog Risk Task (measured at baseline, week 30 and week 56) We will utilize the average number of pumps on un-popped balloons and mean balloons popped.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No